CLINICAL TRIAL: NCT00008203
Title: High-Dose Chemotherapy Followed By Autologous Hematopoietic Stem Cell Support And One Of Two Regimens Aimed At Modifying Immune Reconstitution In Women With High Risk Stage 2 And Stage 3 Breast Cancer
Brief Title: Comparison of Biological Therapies Following Combination Chemotherapy and Bone Marrow or Peripheral Stem Cell Transplantation in Women With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068387; CPMC-IRB-7608; CPMC-CAMP-014; NCI-G00-1890
Record Dates: First submitted 2001-01-06; First posted 2003-06-05 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2003-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — aldesleukin; Interferon-gamma; Carboplatin; Cyclophosphamide; Cyclosporine; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon gamma
Drug: carboplatin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Biological therapy may interfere with the growth of the cancer cells. It is not yet known which post-transplant biological therapy regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of cyclosporine and interferon gamma to that of interleukin-2 following combination chemotherapy and bone marrow or peripheral stem cell transplantation in women who have stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response, disease-free survival (DFS), and overall survival of women with high-risk stage II or III breast cancer treated with high-dose cyclophosphamide, thiotepa, and carboplatin with autologous marrow and/or peripheral blood stem cell transplantation.
* Determine the safety of immunomodulation consisting of cyclosporine and interferon gamma versus low-dose interleukin-2 in this patient population.
* Determine parameters associated with immune activation and autologous graft-versus-host disease.
* Determine which immunomodulation regimen is more efficacious with respect to DSF.

OUTLINE: This is a randomized study. Patients are stratified according to stage (II vs III), age, lymph node status, and inflammatory histology. Patients are randomized to one of two immunomodulation arms.

Autologous harvest of at least 1 million CD34+ cells /kg or 400 million mononuclear cells/kg must be achieved.

All patients receive cyclophosphamide IV continuously and thiotepa IV continuously over 96 hours on days -6 through -3 and carboplatin IV over 5 hours daily on days -6 through -3. Patients undergo autologous bone marrow and/or peripheral blood stem cell transfusion on day 0.

* Arm I: Patients receive cyclosporine IV over 4 hours twice a day, beginning on day 0 and continuing until discharge from the hospital, and interferon gamma subcutaneously (SC) every 2 days on days 7-28.
* Arm II: Patients receive interleukin-2 SC daily for 28 days following recovery of blood counts.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then annually for 5 years.

PROJECTED ACCRUAL: A total of 70 patients (30 with stage II disease and 40 with stage III disease) will be accrued over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage II with at least 10 lymph nodes involved with malignancy OR
  * Stage III (any T3b-T4, N2 or N3, M0)
* Ineligible for other high priority national or institutional study
* No metastasis to brain (confirmed by CT or MRI)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to physiologic 65

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 times normal

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* LVEF at least 45%

Other:

* HIV negative
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 cycles of prior chemotherapy required
* Stage II patients must have completed 4-6 courses of doxorubicin and/or taxol-based adjuvant chemotherapy
* Stage III patients must have achieved complete or partial response to 4-6 courses of doxorubicin and/or taxol-based induction chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-05; Primary Completion 2005-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Vahdat LT, Cohen DJ, Zipin D, Lo KS, Donovan D, Savage D, Tiersten A, Nichols G, Troxel A, Hesdorffer CS. Randomized trial of low-dose interleukin-2 vs cyclosporine A and interferon-gamma after high-dose chemotherapy with peripheral blood progenitor support in women with high-risk primary breast cancer. Bone Marrow Transplant. 2007 Aug;40(3):267-72. doi: 10.1038/sj.bmt.1705692. Epub 2007 Jun 11. PMID 17563739